CLINICAL TRIAL: NCT03840512
Title: A Phase 2a, Open-label, Multicenter, Study to Evaluate the Pharmacokinetic (PK), Safety and Efficacy of Multiple Doses of Cannabidiol for the Prevention of aGVHD After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: An Open Label Study of Multiple Doses of Cannabidiol in the Prevention of Acute Graft-Versus-Host Disease (GVHD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kalytera Therapeutics Israel, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: KAL05
Record Dates: First submitted 2019-02-10; First posted 2019-02-15 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Prevention aGVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral CBD 75 BID (Experimental)
  Interventions: Drug: CBD
- Oral CBD 150 BID (Experimental)
  Interventions: Drug: CBD
- Oral CBD 300 BID (Experimental)
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — CBD + Standard aGVHD prophylaxis calcineurin inhibitor (cyclosporine or tacrolimus) + methotrexate (MTX).
  Subjects transplanted from unrelated donors or from mismatched siblings will also receive anti-T cell globulin.

SUMMARY:
A prospective, open-label, phase 2a study, to evaluate the pharmacokinetic (PK) profile, safety, and efficacy of multiple doses of Cannabidiol (CBD) in participants Graft-Versus-Host Disease (GVHD) after allogeneic hematopoietic stem cell transplantation (HSCT)

DETAILED DESCRIPTION:
The study contains 3 cohorts of 12 participants each: All participants will be orally administered for 105 days with CBD at doses of 75, 150 or 300 mg (PO) BID for the prevention of acute GVHD (aGVHD) following allogeneic HSCT.

In addition to the study drug, all participants will receive standard aGVHD prophylaxis consisting of a calcineurin inhibitor (cyclosporine or tacrolimus) and a short course of methotrexate (MTX). After completion of 105 treatment days, the participant will be followed-up until day 180.

ELIGIBILITY:
Inclusion Criteria:

1. Any malignant hematological disease in CR or Myelodysplastic Syndrome (MDS)
2. Age ≥ 18 years
3. Karnofsky Score (KS) ≥ 60%
4. HSCT-Comorbidity Index (HSCT-CI) score ≤ 3
5. No major organ dysfunction
6. Myeloablative or reduced intensity conditioning regimen
7. Matched (7/8 or 8/8) unrelated donor
8. Peripheral blood stem cell graft
9. Female subjects of childbearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for the follow-up time period. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
10. Male subjects with partners of childbearing potential must agree to use adequate contraception (barrier method or abstinence) during the study.
11. Subject's written informed consent

Exclusion Criteria:

1. Malignant hematological disease other than MDS, not in CR
2. Myelofibrosis
3. Allogeneic transplantation from a matched or mismatched sibling donor
4. Cord blood transplantation
5. Positive serology for HIV
6. Serious psychiatric or psychological disorders
7. Any uncontrolled infection at time of registration
8. Active consumption of illicit drugs (such as: Crack cocaine, Heroin, Methamphetamines, Cocaine, Bath Salts, Amphetamines, Methadone, Benzodiazepine, Ecstasy)
9. Use of Cannabis and/or its derivatives fourteen days prior to HSCT and for the duration of study participation
10. Uncontrolled hepatitis B or active hepatitis C infection.
11. QTc>450ms per Fridericia's correction and Impaired cardiac function or clinically significant cardiac diseases
12. Inadequate renal function defined as measured creatinine clearance > 2.0 mg/dl
13. Liver enzymes: ALT and AST > 3x upper limit of normal
14. Pregnancy or breastfeeding ((positive serum β-HCG 7 days before first dose)
15. Treatment with another investigational drug, biological agent, or device within 30 days of first dose, or investigational cell therapy within 6 months of first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and serious adverse events (SAEs) Reporting | Up to day 180
  All AEs will be recorded, whether considered minor or serious, drug-related or not
Cumulative incidence of aGVHD at day 100 post-transplant | First 100 days after transplant
  Cumulative Incidence of Grade B-D aGvHD
Pharmacokinetic parameters of Cannabidiol (CBD) - Cmax | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile - Cmax - Maximum Plasma Concentration
Pharmacokinetic parameters of Cannabidiol (CBD) - Tmax | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile - Tmax - time to reach maximum plasma concentration
Pharmacokinetic parameters of Cannabidiol (CBD) - Tlag | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile - Tlag - Absorption lag-time defined as the time of the first concentration ≥ Limit of Quantitation (LOQ)
Pharmacokinetic parameters of Cannabidiol (CBD) - AUC0-t | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile - AUC0-t - area under the plasma concentration-time curve (AUC0-t) up to the last quantifiable concentration (LOQ) from time of administration (t=0) up to the selected
Pharmacokinetic parameters of Cannabidiol (CBD) - λz | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile: λz - Elimination rate constant determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve
Pharmacokinetic parameters of Cannabidiol (CBD) - T1/2 | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile: T1/2 - Terminal elimination half-life
Pharmacokinetic parameters of Cannabidiol (CBD) - AUC0-∞ | Blood samples will be obtained on Day 7 before HSCT and Day 7 post HSCT. Sampling times: immediately after CBD dosing and at 15, 30, 45, 60, 120, 180, and 240 minutes, and 8, 12 and 24 hours after dosing of CBD
  Pharmacokinetic (PK) profile: AUC0-∞ - area under the plasma concentration-time curve extrapolated to infinity
Cumulative incidence of aGVHD at day 180 post-transplant | Day 180 post-transplant
  Cumulative Incidence of Grade 2-4 aGvHD

CONTACTS AND LOCATIONS:
Locations (5):
- St Vincent's Hospital Sydney - The Kinghorn Cancer Centre, Sydney, Australia
- Israel (4):
  - Rambam Health Care - Bone Marrow Transplantation Unit, Haifa
  - Hadassah Medical Center - Bone Marrow Transplantation Department, Cancer Immunotherapy and Immunobiology Research Center, Jerusalem
  - Davidof Cancer Center, Beilinson hospital, Rabin medical center, Petah Tikva
  - Tel-Aviv Sourasky Medical Center - Bone Marrow Transplantation Unit, Tel Aviv